CLINICAL TRIAL: NCT04291690
Title: The TARGET-EFT Trial (MulTicomponent Acute Intervention in FRail GEriatric PaTients With Cardiovascular Disease Using the Essential Frailty Toolset)
Brief Title: The TARGET-EFT Randomized Clinical Trial
Acronym: TARGET-EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Afilalo (Other)
Responsible Party: Sponsor-Investigator, Jonathan Afilalo, Director, Geriatric Cardiology Fellowship Program, Division of Cardiology and Centre for Clinical Epidemiology, Jewish General Hospital, McGill University, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TARGET-EFT 2020-2077
Record Dates: First submitted 2020-01-09; First posted 2020-03-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Frailty; Cardiovascular Diseases in Old Age; Geriatric Cardiology; Quality of Life
Keywords: Randomized Clinical Trial; Frailty; Intervention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Single-center randomized clinical trial with parallel group design at the Jewish General Hospital (JGH); an academic tertiary care center in Montreal, Quebec, Canada.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the allocated group of the patients, and they will not be the same team members that delivered the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Usual clinical care as prescribed by their treating clinicians; which may or may not include physiotherapy, geriatric consultation, nutritional consultation and supplementation, and treatment of anemia.
- Intervention Group (Experimental): Multi-component intervention in addition to usual care; which may include - in a targeted fashion - physical training for those with physical weakness, cognitive stimulation for those with cognitive impairment, oral nutritional supplementation for those with malnutrition, and intravenous iron replacement therapy for those with iron deficiency anemia.
  Interventions: Other: Physical Component of the Intervention; Other: Cognitive Component of the Intervention; Other: Nutritional Component of the Intervention; Other: Iron-Deficiency Anemia (IDA) Component of the Intervention

INTERVENTIONS:
Other: Physical Component of the Intervention — We will encourage and assist patients to walk around the ward as tolerated and approved by their treating clinicians, to maximize the time spent out of bed, minimize the time spent in bed, and to encourage and assist them to perform chair rises to build lower extremity strength. For selected intervention patients with greater physical weakness, defined as SPPB ≤9, a Certified Exercise Physiologist will administer a supervised multicomponent exercise program combining strength, flexibility, balance and gait for the prevention of weakness and falls. The exercise program is adapted from the Vivifrail program which is an EU-funded initiative that provides a guide to prevent frailty, physical deconditioning, and incident disability in older persons. The program includes two daily sessions, one in the morning and one in the afternoon, for a duration of 20 minutes each. The morning session includes strength and flexibility exercises. The afternoon session targets balance and walking.
  Arms: Intervention Group
Other: Cognitive Component of the Intervention — We will encourage and assist them to wear their hearing and visual aids (if they have these), orient them to time and place verbally and in writing on a clearly visible white-board in their hospital room - and also encourage their family members and caregivers to do so on a regular basis, and inquire about their sleep quality and communicate with the clinical team to reduce sleep disturbances. For selected intervention patients with greater cognitive impairments, defined as MMSE ≤26, we will provide cognitive simulation twice daily during the scheduled visits. Cognitive stimulation comprises of activities with the patient, including but not limited to current news, trivia, crossword puzzles, and memory games. These cognitive interventions are adapted from the Hospital Elder Life Program (HELP) that targets risk factors for delirium.
  Arms: Intervention Group
Other: Nutritional Component of the Intervention — We will reinforce proper eating habits, encourage and assist patients to wear their dentures (if they have these), and inquire about their food preferences and eating barriers and communicate with the clinical dieticians to address these issues. For selected intervention patients with greater nutritional deficits, defined as a positive PONS, we will recommend to the treating clinicians to prescribe MedPass supplementation. PONS, developed as a preoperative screening tool but also used in nonoperative medical settings, reflects low body mass index, weight loss, low dietary intake, and albumin level. MedPass is a 60 mL calorically dense (2 kcal/mL) oral nutritional supplement consumed between meals 4 times per daily. If MedPass supplementation is contraindicated, the treating team will have the full discretion not to prescribe it and/or to consider alternative supplementation strategies.
  Arms: Intervention Group
Other: Iron-Deficiency Anemia (IDA) Component of the Intervention — We will verify their clinical blood test results for hemoglobin level and iron studies and apply the diagnostic criteria for iron deficiency as recommended by the Canadian Cardiovascular Society Guidelines for Heart Failure. These criteria are: (i) Hemoglobin <130g/L in men or <120g/L in women with (ii) a Ferritin <100μg/L or a Ferritin <300μg/L with a Saturation <20%. For selected intervention patients with diagnosed iron deficiency anemia, according to these established criteria, we will recommend to the treating clinicians to prescribe Venofer intravenous iron replacement therapy. The use of intravenous iron replacement therapy is a Strong Recommendation in the Canadian Cardiovascular Society Guidelines. Venofer is prescribed at a dosage of 300 mg IV daily for a total of 3 doses. If Venofer supplementation is contraindicated, the treating team will have the full discretion not to prescribe it and/or to consider alternative strategies.
  Arms: Intervention Group

SUMMARY:
Randomized clinical trial to determine whether a multicomponent intervention will lead to improvements in mobility, self-care, mood, pain, and physical activity among frail and pre-frail older adults (as measured with the Essential Frailty Toolset; EFT) hospitalized for an acute cardiovascular illness.

DETAILED DESCRIPTION:
The investigators will conduct a single-center randomized clinical trial at the Jewish General Hospital; an academic tertiary care center in Montreal, Quebec. Researchers will pre-screen stable patients ≥65 years of age admitted to the cardiovascular unit. The investigators will target those that consent and have evidence of frailty or pre-frailty according to the EFT (score ≥1/5). The EFT consists of a chair rise test to screen for physical frailty, a mini-cog test to screen for cognitive impairment, a hemoglobin level and a serum albumin level. Patients will be randomly allocated to the usual-care control group, or the intervention group that will receive targeted treatments depending on the EFT deficits identified. All patients will be outfitted with a hip-worn accelerometer to monitor position, step count, and sleep data during the study period. Patients will undergo a structured questionnaire and physical performance assessment at baseline (upon index admission) and at discharge, and will be contacted by telephone 30 days post-discharge to assess their recovery. The primary endpoint will be represented by the EQ-5D scale (mobility, self-care, mood, pain, and physical activity) measured by blinded observers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Frail or pre-frail as defined by EFT score ≥1
* Admission to the JGH cardiovascular unit
* Signed informed consent

Exclusion Criteria:

* Expected discharge within <3 days
* Clinically unstable (unstable vital signs, low-threshold coronary ischemia, uncontrolled heart failure, uncontrolled arrhythmia)
* Awaiting cardiac surgery during the index hospitalization
* Severe dementia (MMSE ≤10/30)
* Delirium (CAM positive)
* Psychiatric condition precluding cooperation
* Not English or French speaking
* Parkinson's disease
* Recent stroke <7 days
* Bed-bound or paraplegic
* End-of-life care plan

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life: EQ-5D-5L scale | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Self-reported health-related quality of life is measured with EQ-5D at baseline and discharge. Items are scored level 1-5 (1 = no problems, 5 = unable/extreme problems). The visual analog scale is scored 0-100 (0 = worse imaginable health ever, 100 = best imaginable health ever). The scale generates a descriptive set that is compared to value sets to produce a value index.

SECONDARY OUTCOMES:
Change in health-related quality of life: EQ-5D-5L scale | From date of hospital discharge (assessed up to 6-weeks) to 30-days post-discharge (assessed up to 10 weeks)
  Self-reported health-related quality of life is measured with EQ-5D at 30-days post-hospitalization. Items are scored level 1-5 (1 = no problems, 5 = unable/extreme problems). The visual analog scale is scored 0-100 (0 = worse imaginable health ever, 100 = best imaginable health ever). The scale generates a descriptive set that is compared to value sets to produce a value index.
Change in Hospital-Acquired disability | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Hospital-acquired disability will be measured using the Older Americans Resources and Services (OARS) Activities of Daily Living (ADL) Scale. ADLs will be assessed at baseline and discharge. Each item is scored 1-3 (1 = without help, 3 = completely unable to), yielding a total score of 0-7.
Hospital-acquired disability | From date of hospital discharge (assessed up to 6-weeks) to 30-days post-discharge (assessed up to 10 weeks)
  Hospital-acquired disability will be measured using the Older Americans Resources and Services (OARS) Activities of Daily Living (ADL) Scale. ADLs will be assessed at 30-days post-hospitalization. Each item is scored 1-3 (1 = without help, 3 = completely unable to), yielding a total score of 0-7.
Number of participants with all-cause death, delirium, fall, infection, pressure ulcer | Date of randomization until date of first documented progression of all-cause death, delirium, fall, infection, pressure ulcer assessed up to hospital discharge (assessed up to 6-weeks)
  Composite endpoint
Number of participants with all-cause death, discharge to healthcare facility, unplanned repeat hospital visit | Date of hospital discharge (assessed up to 6-weeks) until date of first documented progression of all-cause death, discharge to healthcare facility, unplanned repeat hospital visit assessed up to 30-days from hospital discharge
  Composite endpoint
Length of stay | Date of cardiovascular unit admission to hospital discharge (assessed up to 6-weeks)
  Number of days from cardiovascular unit admission to hospital discharge.
Time out of bed | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Average number of hours per day out of bed recorded by actigraphy
Lower extremity physical performance | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Lower extremity weakness will be assessed using the Short Physical Performance Battery scale (SPPB) at baseline and discharge. SPPB is scored 0-12 (0 = worst physical performance, 12 = best physical performance).

OTHER OUTCOMES:
Frailty | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Frailty will be assessed using the Essential Frailty Toolset (EFT) scale during hospital stay. Each item is scored from 0-2 points, yielding a total score of points 0-5.
Frailty | From date of hospital discharge (assessed up to 6-weeks) to 30-days post-discharge (assessed up to 10 weeks)
  Sarcopenia will be assessed with the SARC-F scale at 30 days post-hospital discharge. Each item is scored 0-2 (0 = none, 2 = a lot or unable), yielding a total score of 0-10.
Mobility | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Mobility during hospital stay will be measured using the Level of Function (LOF) scale. LOF is scored level 0-5 (0 = not responsive, not able to cooperate in care and is bed-bound, 5 = able to tolerate increased distances in walking around the unit).
Change in skeletal muscle mass | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Skeletal muscle mass will be measured using a portable bioimpedance and/or ultrasound devices at baseline and discharge.
Step counts | Date of randomization to hospital discharge (assessed up to 6-weeks)
  Physical activity will be measured during the hospital stay. Average number of steps per day are recorded by actigraphy.
Anxiety and depression | Hospital discharge (assessed up to 6-weeks)
  Self-reported hospital anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS) at discharge. Items scored 0-3 (0 = no sign of anxiety/depression, 3 = signs of extreme anxiety/depression), yielding a total score of 0-21 for anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Afilalo, MD, MSc, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Fountotos R, Ahmad F, Bharaj N, Munir H, Marsala J, Rudski LG, Goldfarb M, Afilalo J. Multicomponent intervention for frail and pre-frail older adults with acute cardiovascular conditions: The TARGET-EFT randomized clinical trial. J Am Geriatr Soc. 2023 May;71(5):1406-1415. doi: 10.1111/jgs.18228. Epub 2023 Jan 16. PMID 36645227